CLINICAL TRIAL: NCT02949323
Title: Etiological Diagnosis of Urinary Stone in Chinese Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hongquan Geng, Director, Department of Pediatric Urology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-026
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Stone
Keywords: children; renal stone; metabolic evaluation; Mutational analysis
MeSH Terms: conditions — Urinary Calculi; Nephrolithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- children with urinary stones: children with urinary stones
  Interventions: Other: urinary stone
- children without urinary stones: children without urinary stones

INTERVENTIONS:
Other: urinary stone — patients of group one have urinary stones
  Groups: children with urinary stones

SUMMARY:
The incidence of nephrolithiasis in children has been reported to increase by approximately 6-10% annually, and the incidence is currently 50 per 100,000 children with high recurrent rate. Investigators aimed to determine the metabolic risk factors in Chinese children through metabolic evaluation.

In order to identify diagnostic criteria of hypocitraturia and hyperoxaluria in western country wether adapt to Chinese children, investigators aim to determine normal urine levels of oxalate and citrate in children without kidney stone.

DETAILED DESCRIPTION:
Investigators aimed to determine the metabolic risk factors in 200 Chinese children with urinary stones through metabolic evaluation.

In order to identify diagnostic criteria of hypocitraturia and hyperoxaluria in western country wether adapt to Chinese children, investigators aim to determine normal urine levels of oxalate and citrate in children without kidney stone.

ELIGIBILITY:
Inclusion Criteria:

* Children with urinary stones

Exclusion Criteria:

* Anatomic urinary system abnormality, vesicoureteral reflux, urinary tract infection (temperature >38°C and/or positive urine culture), solitary kidney, and renal insufficiency

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with urinary stones
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Urinary oxalate; | urine collected in 24 hours

SECONDARY OUTCOMES:
Urinary citrate; | urine collected in 24 hours
Urinary calcium | urine collected in 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hongquan Geng, M.D, Study Chair — Department of Pediatric urology,Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Lei He, M.D, Principal Investigator — Department of Pediatric urology,Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Pediatric urology,Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
no plan